CLINICAL TRIAL: NCT00542048
Title: An Open-label, Uncontrolled, Phase II Trial Evaluating the Single-dose and Steady-state Pharmacokinetics of EndoTAG®-1 and Its Effect on the Blood Supply and the Angiogenesis of Hepatic Metastases in Patients With a Carcinomatous Primary Tumor Other Than Hepatocellular (HCC), Biliary or Bile Duct Carcinoma
Brief Title: A Trial Evaluating the Pharmacokinetics and Mode of Action of EndoTAG®-1 in Tumor Patients With Hepatic Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Dr. Carola Adam/Clinical Project Leader, MediGene
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CT 4003
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2009-11

CONDITIONS: Liver Cancer; Neoplasm Metastasis
Keywords: Hepatic metastases; Angiogenesis; EndoTAG-1; Pharmacokinetics; Pharmacodynamics; Metastases of the liver
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: EndoTAG®-1

INTERVENTIONS:
Drug: EndoTAG®-1 — EndoTAG®-1 22 mg/m² twice weekly

SUMMARY:
The primary objective of study CT 4003 is to assess the behavior of EndoTAG®-1 in the body (making a so-called pharmacokinetic profile). Therefore, the course of the drug in the body is examined, i.e. the amount and speed of the drug uptake as well as the distribution and the elimination of the drug is being investigated. Further objectives of the study are to assess the effect of EndoTAG®-1 on liver metastases concerning size and blood supply measured by imaging techniques (contrast-enhanced ultrasound and magnetic resonance imaging as well as duplex sonography) and to assess the effect on blood markers which are indicators for the destruction and neoplasm of blood vessels (so-called markers of angiogenesis).

DETAILED DESCRIPTION:
Liver metastases are among the most frequent neoplasms of the liver and represent a quite uniform clinical entity regardless from which carcinoma they originate. The treatment is dependent on number and size of the hepatic lesions but still, none of the therapeutic options leads to satisfying results. The growth of tumors and metastases is dependent on blood vessels, which supply the tumors and metastases with nutrients. Liver metastases, independent from which original tumor they come from, are especially well supplied with blood. The aim of the treatment with the investigational medicinal product EndoTAG®-1 is to target the blood vessels, which supply the metastases, and destroy them. Consequently, the metastases themselves will be damaged.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable hepatic metastases of a carcinomatous origin with exception of HCC, biliary or bile duct carcinoma
* At least one measurable hepatic metastases > 20 mm in diameter (measured in MRI)
* Last application of palliative chemotherapy (drug dependent on the primary tumor) at least 7 days ago
* Gender: male and female (at least 6 individuals of each gender)
* Age >= 18 years
* Negative pregnancy test (females of childbearing potential)
* Willingness to perform double-barrier-contraception during the study and for 6 month post study medication
* ECOG performance status 0,1 or 2
* Assumed life expectancy of > 3 month
* Signed informed consent

Exclusion Criteria:

* History of significant liver pathology (other than metastases, e.g. cirrhosis of the liver, PSC, PBC) or liver transplantation
* Laboratory tests (hematology, chemistry) outside specific limits:
* ANC <= 1.0 x 10^9/L
* Platelets <= 100 x 10^9/L
* Hb <= 9.0 g/dL (<= 5.6 mmol/L)
* Total Bilirubin > 2.0 mg/dL
* Serum Creatinine > 1.5 mg/dL
* Renal insufficiency with a GFR < 60 mL/min
* Currently ongoing taxane-containing palliative chemotherapy regimen or history of taxane administration within 4 weeks prior to study entry
* Pregnancy or nursing status
* Positive HIV, HBV or HCV testing
* The patient has a contraindication for MRI or CEUS according to accepted clinical guidelines
* Known hypersensitivity to any component of the EndoTAG®-1 formulation, gadolinium-based MR-contrast media or sulphur hexafluoride
* Claustrophobia or history of active or significant neurological disorder and/or psychiatric disorder that would prohibit the understanding and giving of informed consent, or would interfere in the clinical and radiological evaluation of the patient during the trial
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | Last patient out

SECONDARY OUTCOMES:
Tumor response, Tumor perfusion, Soluble markers of angiogenesis, Pharmacodynamics, Safety | Last patient out

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mross, PD, Principal Investigator — Klinik für Tumorbiologie an der Albert-Ludwigs-Universität Freiburg
Locations (1):
- Klinik für Internistische Onkologie in der KTB Klinik für Tumorbiologie an der Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau, Baden-Würtemberg, Germany